CLINICAL TRIAL: NCT00060918
Title: A Randomized, Double-Blind, Multicenter Study Comparing the Glycemic Control Characteristics of Carvedilol and Metoprolol in Hypertensive Patients With Type II Diabetes Mellitus.
Brief Title: Glycemic Control Of Carvedilol Versus Metoprolol In Patients With Type II Diabetes Mellitus And Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105517/346
Record Dates: First submitted 2003-05-15; First posted 2003-05-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: Type 2 diabetes; hypertension; beta-blockers
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carvedilol
Drug: metoprolol
  Other Names: carvedilol

SUMMARY:
To evaluate the effects of two different antihypertensive medications in the drug class of beta-blockers on control of glucose in Type II diabetic patients with high blood pressure.

ELIGIBILITY:
Inclusion criteria:

* Patients at screening must be insulin producing Type II diabetics (C peptide positive).
* Must have a history of mild to moderate hypertension (140-179 systolic; 90-1-9 diastolic).
* Must be on stable regimen of ACE (angiotensin converting enzyme) / ARB (angiotensin receptor blocker) treatment alone or in combination with other treatments.
* Patient''s laboratory result for HbA1c must be 6.5 - 8.5 (drug treated) or 6.5 - 7.5 (diet alone).
* Must be on a stable antidiabetic regimen (drug treated or diet alone).

Exclusion criteria:

* Patients using beta-blocker therapy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1210
Dates: Start 2001-06; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 5 months | 5 months

SECONDARY OUTCOMES:
Blood pressure at 3 and 5 months. Body weight at 3 and 5 months. Lab values (glucose, insulin, triglycerides, cholesterol, and albumin:creatinine ratio) at 3 and 5 months. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (46):
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Burlingame, California
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Hemet, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Luis Obispo, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, O'Fallon, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Oak Park, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Oregon City, Oregon
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, The Colony, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin